CLINICAL TRIAL: NCT03288142
Title: Improving Hypertension Using a Smartphone-Enabled Personal Control Program: The Smart Hypertension Control Study
Brief Title: The Smart Hypertension Control Study
Acronym: iSmartHyp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Omron Healthcare Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Stephen Persell, MD, MPH, Associate Professor of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STU00205025
Record Dates: First submitted 2017-09-15; First posted 2017-09-19 (Actual); Results first posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with randomization stratified by age and baseline systolic blood pressure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Hypertension Coaching Application and Home Monitor: (Experimental): The intervention group will receive all the interventions provided to the control group. In addition, intervention group participants will install on their mobile phone the hypertension personal control program (HPCP) ("Lark HTN Pro"), which is a smartphone application. The intervention group will have the HPCP installed on their iOS device during their initial office visit (screening/baseline) and will successfully take a reading from their HBMD. The HPCP has blood pressure, medication, and weight monitoring, including periodic reminders for the user to measure blood pressure, measure weight, and take their medication(s). The HPCP provides real-time feedback based on user input, such as out-of-range measurements and has additional features designed to encourage behavior change in areas such as dietary intake, physical activity, sleep, and stress reduction. Users can set goals and receive guidance and feedback through the app.
  Interventions: Other: Hypertension Coaching Application and Home Monitor
- Control:Tracking Application and Home Monitor: (Active Comparator): Control group participants will be provided with a home blood pressure monitoring device (HBMD) (Omron BP761N Bluetooth Smart Automatic Upper Arm Blood Pressure Monitor) and will be instructed in its use at the baseline study visit. Participants will also receive an information sheet describing home blood pressure monitoring that gives advice for how to respond to different home readings. At the baseline visit, participants will be instructed to install an Omron application to their smart phone device (to monitor use of the HBMD). Participants will continue to receive all routine care, including anti-hypertensive medications as prescribed by their regular clinicians.
  Interventions: Other: Control: Tracking Application and Home Monitor

INTERVENTIONS:
Other: Hypertension Coaching Application and Home Monitor — The intervention group will have the HPCP installed on their iOS device during their initial office visit (screening/baseline) and will successfully take a reading from their HBMD
  Other Names: Lark HTN Pro
  Arms: Intervention: Hypertension Coaching Application and Home Monitor:
Other: Control: Tracking Application and Home Monitor — Control group participants will be provided with a home blood pressure monitoring device (HBMD) (Omron BP761N Bluetooth Smart Automatic Upper Arm Blood Pressure Monitor) and will be instructed in its use at the baseline study visit. Participants will also receive an information sheet describing home blood pressure monitoring that gives advice for how to respond to different home readings. At the baseline visit, participants will be instructed to install an Omron application to their smart phone device (to monitor use of the HBMD). Participants will continue to receive all routine care, including anti-hypertensive medications as prescribed by their regular clinicians.
  Arms: Control:Tracking Application and Home Monitor:

SUMMARY:
Investigators at Northwestern University will partner with Omron Healthcare Co., Ltd. (hereinafter referred to as "Omron") to conduct a randomized controlled trial of a hypertension personal control program (HPCP), known as Lark HTN Pro with a home blood pressure monitoring device (HBMD) compared to a HBMD alone. The overarching goal of this study is to investigate the effects of the HPCP on blood pressure, blood pressure self-management behaviors, and healthy lifestyle behaviors among adults with hypertension.

DETAILED DESCRIPTION:
The study team used structured language queries of electronic health record data from the Northwestern Medicine Enterprise Data Warehouse (NMEDW) to identify potentially-eligible participants with elevated blood pressure and exclude patients with clinical exclusion criteria from Northwestern Medical Group outpatient practices. During the on-site visit individuals were asked to provide written informed consent and have blood pressure measured in a standardized fashion to see if this inclusion criteria is met.

We conducted a non-blinded randomized controlled trial among hypertensive adults in NMG outpatient clinics. We randomized participants in a 1:1 fashion to the intervention group (HPCP + HBMD) or the comparator group (HBMD alone). Randomization was performed using a centralized computer-generated assignment sequence uploaded a priori to Northwestern University's REDCap (Research Electronic Data Capture) application. Randomization was stratified by: age (<65 or ≥65 years of age) and baseline systolic blood pressure (<145 or ≥145 mmHg) to optimize the likelihood of obtaining similar populations in each treatment group.

We recruited adults with elevated blood pressure as assessed by in-person standardized examination at baseline. We measured change in blood pressure by in-person examination at 6 months. We recruited between 350 to 400 participants in order to have 333 participants with analyzable data at the time of study completion. If changes were deemed necessary, a revision to the study protocol was submitted to the IRB for review and approval prior to implementing these changes.

Control group participants were provided with a home blood pressure monitoring device (HBMD) (Omron BP761N Bluetooth Smart Automatic Upper Arm Blood Pressure Monitor) and will be instructed in its use at the baseline study visit. Participant also received an information sheet describing home blood pressure monitoring that gives advice for how to respond to different home readings. At the baseline visit, participants were instructed to install an Omron application to their smart phone device (to monitor use of the HBMD). Participants continued to receive all routine care, including anti-hypertensive medications as prescribed by their regular clinicians.

The intervention group received all the interventions provided to the control group. Intervention group participants were sent a hyperlink to install the hypertension personal control program (HPCP) ("Lark HTN Pro"), which is a smartphone application installed on their iOS device during their initial office visit (screening/baseline) and successfully took a reading from their HBMD. The HPCP has blood pressure, medication, and weight monitoring, including periodic reminders for the user to measure blood pressure, measure weight, and take their medication(s). The HPCP provides real-time feedback based on user input, such as out-of-range measurements and has additional features designed to encourage behavior change in areas such as dietary intake, physical activity, sleep, and stress reduction.

Study participants were required to return for a 6-month study visit (within 2 weeks before to 4 weeks after). During the 6-month visit, subjects had their height/weight and blood pressure measured again. Participants also repeated questionnaires related to their current cardiovascular medications. They also completed questionnaires measuring: medication adherence, self-efficacy, diet, physical activity, and sleep duration. An exit survey was provided to participants at the end of the 6-month follow up visit to obtain feedback on Lark and Omron apps usability.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years to <85 years at the time of screening
* Standardized mean blood pressure measurement ≥135 to <180 mmHg systolic or ≥85 to <110 mmHg diastolic
* Have and use an iOS device(s) (iPhone generation 5s or newer)
* Able to provide written informed consent prior to participation in the study
* Receive their primary care from a Northwestern Medicine clinic site

Exclusion Criteria:

* Current user of the HCPC (Lark HTN Pro)
* Standardized mean blood pressure measurement ≥180 mmHg systolic or ≥110 mmHg diastolic
* Persistent atrial fibrillation as indicated in the electronic health record (EHR)
* Pregnant or planning to become pregnant during the study period
* Severe kidney disease, defined as estimated glomerular filtration rate <30 per 1.73 m2 or currently on renal replacement therapy (i.e. hemodialysis or peritoneal dialysis)
* Hearing impaired and unable to respond to phone calls
* Lack of fluency in English
* History of a cardiovascular event (stroke, transient ischemic attack, myocardial infarction, coronary artery bypass grafting) in the past 3 months
* Diagnosis of dementia as indicated in the electronic health record
* Diagnosis of psychosis as indicated in the electronic health record
* Terminal cancer diagnosis or NYHA III or IV heart failure
* Deemed unsuitable for study by primary care provider
* Individuals requiring BP monitor cuff size larger than 17 inches or 42cm

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2019-04-28 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Persell, MD/MPH, Principal Investigator — Northwestern Medicine
Locations (1):
- Northwestern Medical Group, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Persell SD, Peprah YA, Lipiszko D, Lee JY, Li JJ, Ciolino JD, Karmali KN, Sato H. Effect of Home Blood Pressure Monitoring via a Smartphone Hypertension Coaching Application or Tracking Application on Adults With Uncontrolled Hypertension: A Randomized Clinical Trial. JAMA Netw Open. 2020 Mar 2;3(3):e200255. doi: 10.1001/jamanetworkopen.2020.0255. PMID 32119093

RESULTS

PARTICIPANT FLOW:
Groups:
- Hypertension Coaching Application and Home Monitor: The intervention group will receive all the interventions provided to the control group. In addition, intervention group participants will install on their mobile phone the hypertension personal control program (HPCP) ("Lark HTN Pro"), which is a smartphone application. The intervention group will have the HPCP installed on their iOS device during their initial office visit (screening/baseline) and will successfully take a reading from their HBMD. The HPCP has blood pressure, medication, and weight monitoring, including periodic reminders for the user to measure blood pressure, measure weight, and take their medication(s). The HPCP provides real-time feedback based on user input, such as out-of-range measurements and has additional features designed to encourage behavior change in areas such as dietary intake, physical activity, sleep, and stress reduction. Users can set goals and receive guidance and feedback through the app.
- Tracking Application and Home Monitor: Control group participants will be provided with a home blood pressure monitoring device (HBMD) (Omron BP761N Bluetooth Smart Automatic Upper Arm Blood Pressure Monitor) and will be instructed in its use at the baseline study visit. Participants will also receive an information sheet describing home blood pressure monitoring that gives advice for how to respond to different home readings. At the baseline visit, participants will be instructed to install an Omron application to their smart phone device (to monitor use of the HBMD). Participants will continue to receive all routine care, including anti-hypertensive medications as prescribed by their regular clinicians.
Period: Overall Study
Arm/Group | Hypertension Coaching Application and Home Monitor | Tracking Application and Home Monitor
Started | 166 | 167
Completed | 144 | 152
Not Completed | 22 | 15
Not completed — Lost to Follow-up | 22 | 15

BASELINE CHARACTERISTICS:
Population: 166 participants contributed data for the hypertension coaching application arm of the study. 167 participants from the tracking application arm contributed data to the study. Overall number of participants is 333. 22 participants from intervention arm were excluded from analyses for various reasons leaving 144 participants for analyses.1 missing data and 14 participants were lost to follow up and were excluded from analyses in the control arm which leaves us with 153 participants for analyses.
Groups:
- Hypertension Coaching Application and Home Monitor: Arm assigned hypertension coaching application and home monitor
- Tracking Application and Home Monitor: Arm assigned tracking application and home monitor
- Total: Total of all reporting groups
Arm/Group | Hypertension Coaching Application and Home Monitor | Tracking Application and Home Monitor | Total
Number analyzed (Participants) | 144 | 152 | 296
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 22 participants from intervention arm were excluded from analyses for various reasons.14 participants were lost to follow up and were excluded from analyses in the control arm.
  years | 59.6 (12.4) | 58.3 (13.2) | 58.9 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 22 participants from intervention arm were excluded from analyses for various reasons. 14 participants were lost to follow up and were excluded from analyses in the control arm.
  Participants
    Female | 91 | 91 | 182
    Male | 53 | 61 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 22 participants from intervention arm were excluded from analyses for various reasons. 14 participants were lost to follow up and were excluded from analyses in the control arm.
  Participants
    Hispanic or Latino | 10 | 13 | 23
    Not Hispanic or Latino | 134 | 139 | 273
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 22 participants from intervention arm were excluded from analyses for various reasons. 14 participants were lost to follow up and were excluded from analyses in the control arm.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 4 | 9 | 13
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 56 | 47 | 103
    White | 73 | 79 | 152
    More than one race | 11 | 17 | 28
    Unknown or Not Reported | 0 | 0 | 0
Education [Count of Participants; unit: Participants] — Population: 22 participants from intervention arm were excluded from analyses for various reasons. 14 participants were lost to follow up and were excluded from analyses in the control arm.
  Participants
    Less thank HS graduate | 3 | 2 | 5
    Grade 12 or GED | 10 | 16 | 26
    College 1-3y | 27 | 28 | 55
    College≥4 | 103 | 106 | 209
    Unknown | 1 | 0 | 1
Primary Language [Count of Participants; unit: Participants] — Population: 22 participants from intervention arm were excluded from analyses for various reasons. 14 participants were lost to follow up and participants were excluded from analyses in the control arm.
  Participants
    English | 141 | 143 | 284
    Other | 3 | 8 | 11
    Refused | 0 | 1 | 1
No. of antihypertensive agents used [Count of Participants; unit: Participants] — Population: 22 participants from intervention arm were excluded from analyses for various reasons. 14 participants were lost to follow up and were excluded from analyses in the control arm.
  Participants
    0 | 34 | 53 | 87
    1 | 61 | 44 | 105
    2 | 35 | 40 | 75
    ≥3 | 14 | 15 | 29
Body mass index [Mean (Standard Deviation); unit: kg/m^2] — weight in kilograms divided by height in meters squared. Population: 22 participants from intervention arm were excluded from analyses for various reasons. 14 participants were lost to follow up and were excluded from analyses in the control arm.
  kg/m^2 | 31.9 (8.3) | 31.7 (7.8) | 31.8 (8.0)

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure at 6 Months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmHG
Groups:
- Control: Control group participants will be provided with a home blood pressure monitoring device (HBMD) (Omron BP761N Bluetooth Smart Automatic Upper Arm Blood Pressure Monitor) and will be instructed in its use at the baseline study visit. Participants will also receive an information sheet describing home blood pressure monitoring that gives advice for how to respond to different home readings. At the baseline visit, participants will be instructed to install an Omron application to their smart phone device (to monitor use of the HBMD). Participants will continue to receive all routine care, including anti-hypertensive medications as prescribed by their regular clinicians.
- Intervention: The intervention group will receive all the interventions provided to the control group. In addition, intervention group participants will install on their mobile phone the hypertension personal control program (HPCP) ("Lark HTN Pro"), which is a smartphone application. The intervention group will have the HPCP installed on their iOS device during their initial office visit (screening/baseline) and will successfully take a reading from their HBMD. The HPCP has blood pressure, medication, and weight monitoring, including periodic reminders for the user to measure blood pressure, measure weight, and take their medication(s). The HPCP provides real-time feedback based on user input, such as out-of-range measurements and has additional features designed to encourage behavior change in areas such as dietary intake, physical activity, sleep, and stress reduction. Users can set goals and receive guidance and feedback through the app.
  Lark HTN Pro: The intervention group will have the HPCP
Arm/Group | Control | Intervention
Number analyzed (Participants) | 144 | 152
mmHG
  Systolic BP | 135.0 (13.9) | 132.3 (15.0)
  Diastolic BP | 85.6 (9.8) | 85.1 (9.6)

2. Primary Outcome: Blood Pressure <140/90mmHg
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 144 | 152
Participants | 72 | 78

3. Secondary Outcome: Number of Antihypertensive Agents Used
Description: Number of self reported antihypertensive medication drug classes taken
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Antihypertensives
Arm/Group | Intervention | Control
Number analyzed (Participants) | 144 | 152
Antihypertensives | 1.3 (1.0) | 1.3 (1.2)

4. Secondary Outcome: Antihypertensive Medication Intensification, No. of Additions, Dose Increases, or Substitutions
Description: Number of antihypertensive drug classes that were increased, added or substituted for another drug class
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Antihypertensives
Arm/Group | Intervention | Control
Number analyzed (Participants) | 144 | 152
Antihypertensives | 0.3 (0.6) | 0.4 (0.8)

5. Secondary Outcome: Number of Health System Contacts (Telephone, Office, or Mychart Encounters)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: calls
Arm/Group | Intervention | Control
Number analyzed (Participants) | 144 | 152
calls | 7.0 (11.5) | 6.7 (6.5)

6. Secondary Outcome: Frequency of Home Blood Pressure Measurements Per Month
Description: Frequency of home blood pressure measurements per month derived from home blood pressure monitor for months when home monitoring occurred
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: measurements per month
Arm/Group | Intervention | Control
Number analyzed (Participants) | 144 | 152
measurements per month | 16 [8.5 to 29] | 17 [9 to 32.5]

7. Secondary Outcome: Months When a Home Blood Pressure Reading is Obtained, No.
Description: Number of months out of the 6 month study period when at least one home blood pressure reading was obtained
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Intervention | Control
Number analyzed (Participants) | 144 | 152
Months | 4.9 (1.8) | 5.0 (1.8)

8. Secondary Outcome: Self-efficacy: Confidence in Controlling High Blood Pressure
Description: Self reported response to :How confident are you that you will be able to get your blood pressure controlled and keep it there during the next few months? Reponses were on a 5-point scale ranging from (1) not at all confident to (5) extremely confident.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 144 | 152
units on a scale
  Confidence in controlling blood pressure | 4.4 (0.8) | 4.1 (0.9)
  Confidence in using home monitor | 4.8 (0.6) | 4.7 (0.7)
  Confidence in judging when medication change needed | 4.0 (1.3) | 4.0 (1.2)
  Confidence in doing nonmedication behaviors to control blood pressure | 4.4 (0.9) | 4.4 (0.9)

9. Secondary Outcome: BMI
Description: Body mass index is calculated as the weight in kilograms divided by height in meters squared.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Intervention | Control
Number analyzed (Participants) | 144 | 152
kg/m^2 | 32.0 (8.2) | 31.9 (7.7)

10. Secondary Outcome: Diet Quality Score (as Assessed by Dietary Approaches to Stop Hypertension Questionnaire, DASH-Q
Description: Sum of responses represents intake of foods associated with the Dietary Approaches to Stop Hypertension diet. Range is from 0 to 77 with a higher score indicating better diet. Scores 32 and below indicate a low-quality diet, scores 33 to 51 indicate a medium-quality diet, and scores greater than or equal to 52 indicate a high-quality diet.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 144 | 152
scores on a scale
  Dietary Approaches to Stop Hypertension-Questionnaire score | 38.7 (12.1) | 39.3 (11.8)
  Consumption of processed meats, d/wk | 1.3 (1.6) | 1.5 (1.8)
  Consumption of fried foods, d/wk | 1.0 (1.3) | 1.1 (1.4)
  Consumption of sugar-sweetened beverages, d/wk | 1.7 (2.5) | 1.7 (2.4)
  Consumption of candy, baked goods, or ice cream, d/wk | 2.9 (2.3) | 2.9 (2.2)

11. Secondary Outcome: Minutes Per Week of Self-reported Physical Activity
Description: Self-reported physical activity in minutes per week of at least moderate exercise
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: minutes/week
Arm/Group | Intervention | Control
Number analyzed (Participants) | 144 | 152
minutes/week | 177.6 (169.2) | 143.1 (156.4)

12. Secondary Outcome: Self-reported Sleep Duration
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: sleep hours
Arm/Group | Intervention | Control
Number analyzed (Participants) | 144 | 152
sleep hours | 6.6 (1.4) | 6.5 (1.2)

ADVERSE EVENTS:
Time Frame: 1 year
Description: We assessed adverse events for the duration of the duration of the study. We are not aware of any serious adverse events or deaths and had no events reported to study personnel during the study period. Because no adverse events were reported, we noted this in the required section but want readers to be aware that adverse events were not retorted by any participant to study team.
Groups:
- Intervention: The intervention group will receive all the interventions provided to the control group. In addition, intervention group participants will install on their mobile phone the hypertension personal control program (HPCP) ("Lark HTN Pro"), which is a smartphone application. The intervention group will have the HPCP installed on their iOS device during their initial office visit (screening/baseline) and will successfully take a reading from their HBMD. The HPCP has blood pressure, medication, and weight monitoring, including periodic reminders for the user to measure blood pressure, measure weight, and take their medication(s). The HPCP provides real-time feedback based on user input, such as out-of-range measurements and has additional features designed to encourage behavior change in areas such as dietary intake, physical activity, sleep, and stress reduction. Users can set goals and receive guidance and feedback through the app.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/166 | 0/167
Serious Adverse Events (participants affected / at risk) | 0/166 | 0/167
Other Adverse Events (participants affected / at risk) | 0/166 | 0/167

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/42/NCT03288142/Prot_SAP_000.pdf